CLINICAL TRIAL: NCT05586100
Title: Neoadjuvant and Adjuvant Toripalimab and Cetuximab in Patients With Recurrent, Resectable Squamous Cell Carcinoma of Head and Neck: a Prospective, Single-arm,Phase II Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, ren guoxin, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH9H-2022-T244-1
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Patients With Locally Recurrent Resectable Head and Neck Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cetuximab in combination with toripalimab (Experimental): Participants receive toripalimab administered by intravenous drip at a fixed dose of 240 mg for subjects weighing <50 kg at baseline, using 3 mg/kg. administered every 3 weeks, 2 preoperative and 6 postoperative doses.
  The starting dose of cetuximab is 400 mg/m2, with a titration time of 120 min, and the titration rate should be controlled within 5 ml/min. The maintenance dose is 250 mg/m2 administered weekly for a total of 6 preoperative doses; patients with positive intraoperative pathological margins/extra lymph node envelope invasion are treated with an additional 6 cycles of postoperative cetuximab adjuvant therapy.
  Interventions: Drug: Toripalimab+cetuximab

INTERVENTIONS:
Drug: Toripalimab+cetuximab — Toripalimab administered by intravenous drip at a fixed dose of 240 mg for subjects weighing <50 kg at baseline, using 3 mg/kg. administered every 3 weeks, 2 preoperative and 6 postoperative doses.
  The starting dose of cetuximab is 400 mg/m2, with a titration time of 120 min, and the titration rate should be controlled within 5 ml/min. The maintenance dose is 250 mg/m2 administered weekly for a total of 6 preoperative doses; patients with positive intraoperative pathological margins/extra lymph node envelope invasion are treated with an additional 6 cycles of postoperative cetuximab adjuvant therapy.

SUMMARY:
This study is the first clinical study of Neoadjuvant and Adjuvant treatment of head and neck squamous cell carcinoma with drugs targeting EGFR signaling pathway combined with PD-1 inhibitors, which explores the new combination therapies urgently needed in clinical practice and lays a foundation for subsequent studies, with important scientific research significance and clinical value.

DETAILED DESCRIPTION:
Head and neck cancer is the sixth most common cancer in the world, with more than 550,000 incidences and 300,000 deaths worldwide each year. more than 95% of head and neck cancers are squamous cell carcinomas, and head and neck squamous cell carcinoma (HNSCC) damages and affects patients' appearance and basic physiological, sensory and speech functions, thereby affecting their quality of life. This affects the quality of life of patients. Due to the difficulty of early detection, more than 60% of head and neck squamous cell carcinoma patients are found to be locally advanced, and the prognosis of locally advanced head and neck cancer is poor, with up to 60% of patients experiencing local recurrence and distant metastasis.

Currently, the preferred treatment option for patients with locally recurrent resectable HNSCC is to undergo salvage surgery with or without postoperative local radiotherapy based on pathology, staging, and history of prior radiotherapy. However, even after receiving aggressive treatment, at least 20% of patients with HNSCC still develop local recurrence or distant metastases. In previous studies, the five-year survival rates of patients with locally recurrent, resectable head and neck squamous carcinoma who underwent salvage surgery ranged from 11% to 40%. How to improve the prognosis of patients with locally recurrent, resectable HNSCC is an urgent clinical problem.

The epidermal growth factor receptor (EGFR) is highly expressed in 90% of HNSCC, and high expression of EGFR protein and high copy number of its gene are significantly associated with poor prognosis, short survival, and increased risk of metastasis in HNSCC. The chimeric EGFR-blocking monoclonal antibody cetuximab is approved by the FDA for the first/second-line treatment of recurrent/metastatic, unresectable HNSCC and significantly improves long-term survival in recurrent/metastatic, unresectable HNSCC compared with chemotherapy alone. In the 2021 edition of the CSCO guidelines, cetuximab is recommended as a Class I expert in combination with chemotherapy for the first-line treatment of recurrent/metastatic HNSCC without indications for surgery and radiotherapy (Class 1A evidence), and as a Class II expert in single-agent use for the second-line or salvage treatment of recurrent/metastatic HNSCC without indications for surgery and radiotherapy (Class 2A evidence). Meanwhile, it was approved by the CFDA in February 2020 in combination with platinum and fluorouracil chemotherapy for the first-line treatment of recurrent/metastatic HNSCC, and was successfully covered by Medicare in November 2021. However, whether cetuximab provides a survival benefit in patients with locally recurrent, resectable HNSCC has not been reported in studies.

The successful development of programmed death receptor 1 (PD-1) immune checkpoint inhibitors has significantly impacted the treatment of HNSCC. In patients with unresectable recurrent or metastatic HNSCC resistant to platinum-based therapy, KEYNOTE-040 compared pembrolizumab with the investigator's choice of treatment regimen (docetaxel, methotrexate, or cetuximab), and this trial was just short of the primary endpoint (improved overall survival with pembrolizumab) in the intention-to-treat population (8.4 months in the pembrolizumab group [95% CI, 6.4 to 9.4] vs. 6.9 months [95% CI, 5.9 to 8.0] in the standard treatment group; hazard ratio for death, 0.80; 95% CI, 0.65 to 0.98; P=0.02). In the CheckMate 141 trial, which randomized patients who had received prior platinum-based therapy in a 2:1 ratio to receive either nivolumab or a regimen of the investigator's choice, respectively. Nivolumab improved overall survival (7.5 months [95% CI, 5.5 to 9.1] vs. 5.1 months [95% CI, 4.0 to 6.0]; hazard ratio for death, 0.70; 97.73% CI, 0.51 to 0.96; P=0.01), remission rate (13.3% vs. 5.8%) and 6-month progression-free survival (19.7% vs. 9.9%), and reduced the incidence of serious adverse events (13.1% vs. 35.1%). After more than 2 years of follow-up, a survival benefit of nivolumab treatment remained for patients (hazard ratio for death, 0.68; 95% CI, 0.54 to 0.86; 24-month overall survival, 16.9% vs. 6.0%). The U.S. Food and Drug Administration (FDA) approved both pembrolizumab and nivolumab in 2016 for second-line treatment of advanced HNSCC because they enabled patients to achieve durable remissions and improved survival. In the KEYNOTE-048 study, 882 patients with previously untreated recurrent or metastatic HNSCC were randomized to receive either pembrolizumab monotherapy, Pembrolizumab + chemotherapy (fluorouracil and platinum-based agents) or the standard treatment regimen of fluorouracil and platinum-based agents + cetuximab (the regimen in the EXTREME trial), which confirmed that In the first-line treatment of patients with unresectable recurrent or metastatic HNSCC, pembrolizumab combined with chemotherapy significantly improved overall survival in the total population, and pembrolizumab alone in those with CPS ≥ 1, compared with the traditional EXTREME regimen of targeted chemotherapy, and the FDA approved pembrolizumab for the first-line treatment of advanced HNSCC in 2019.

Currently, immunotherapy and EGFR-targeted therapy for combination therapy have been explored in several studies. The basic rationale supporting these combination therapies is that the two therapies combine different immunological and tumor biological mechanisms that enhance antitumor activity; it is well known that anti-PD-1 therapy enhances cytotoxic T lymphocytes and promotes tumor regression and immune rejection. In contrast, anti-EGFR antibodies induce antibody-dependent cytotoxicity and lead to interactions between immune cells (including natural killer cells and dendritic cells). This interaction can stimulate tumor antigen-specific cellular immunity and generate antigen-specific T-lymphocyte responses [12]. Thus, the two classes of drugs may produce antitumor synergistic effects. In an open-label, multicenter, multicohort phase II clinical trial, the application of pembrolizumab in combination with cetuximab in 33 patients with unresectable recurrent/metastatic HNSCC not previously treated with pembrolizumab and cetuximab showed an overall response rate of 45% at 6 months, while the median duration of remission in patients with effective treatment reached 13.3 months, and two other cohorts are currently recruiting and results have not yet been published, initially showing that the combination of immunotherapy and EGFR-targeted therapy holds promise in patients with relapsed/metastatic HNSCC. However, this treatment modality has not been explored in patients with relapsed resectable HNSCC.

In an open-label, multicenter, single-arm phase II clinical trial, patients with locally relapsed resectable HNSCC were treated with the PD-1 inhibitor nivolumab and the NK cell surface molecule KIR inhibitor Lirilumab in a double-exemption study that was expected to enroll 54 patients, but only 28 subjects were ultimately enrolled due to discontinuation of Lirilumab supply. The study found that the enrolled patients achieved a pathological remission rate of 43%, a one-year DFS of 55.2%, and a 2-year DFS rate of 64% and a 2-year OS rate of 80% in subjects who achieved pathological remission, possibly limited by study discontinuation of enrollment, which has shown good long-term efficacy although the primary study endpoint was not met.

JS001 or toripalimab, the most leading investigational drug of Juniper Biologics against various malignancies, is a recombinant humanized anti-PD-1 injectable monoclonal antibody that was approved for marketing by the State Drug Administration (NMPA) of China on December 17, 2018.JS001 has a high binding affinity and can better compete with PD-L1 and PD-L2 binding competition on tumor cells, while inducing endocytosis of PD-1 receptors and reducing PD-1 expression on the cell membrane surface. Results from completed clinical trials of toripalimab in a variety of cancers, including malignant melanoma, nasopharyngeal carcinoma, and esophageal squamous cell carcinoma, showed that immune-related adverse events were rare and received the first global conditional approval in China on December 17, 2018, for the treatment of unresectable or metastatic melanoma that was previously unavailable for systemic therapy. Individual cases have shown excellent responsiveness and good tolerability of the combination of toripalimab and single-agent chemotherapy in the first-line treatment of elderly R/M HNSCC, while its therapeutic role in R/M HNSCC remains to be investigated.

Therefore, based on the data of previously reported studies of EGFR-targeted therapy combined with immunotherapy in patients with unresectable recurrent/metastatic HNSCC and the preliminary results of PD-1 combined with KIR inhibitors in patients with locally recurrent resectable HNSCC treated with double-free neoadjuvant therapy, we hypothesized that cetuximab in combination with toripalimab prior to salvage surgery could benefit to this high-risk population of patients with locally recurrent resectable HNSCC. This study is the first clinical study of EGFR-targeted therapy combined with PD-1 inhibitor for the neoadjuvant treatment of locally recurrent resectable HNSCC in China, which is of great scientific significance and clinical value in exploring the urgent need for new combination therapies and new treatment options for this high-risk group of patients with locally recurrent resectable HNSCC, and laying the foundation for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years old, regardless of gender
2. histologically or cytologically confirmed and surgically curable recurrent localized squamous carcinoma of the head and neck (tumor primary sites are oropharynx, oral cavity, hypopharynx, and larynx) without any antitumor systemic therapy during the recurrent stage (allowed as part of treatment for locally advanced tumors and requiring more than 6 months between the end of treatment and the signing of the informed consent)
3. an ECOG score of 0 or 1.
4. an expected survival of ≥ 12 weeks.
5. have at least one measurable lesion according to RECIST 1.1 criteria, and a previously treated lesion with radiation therapy, if disease progression has occurred, may also be a measurable lesion.
6. availability of tumor tissue for PD-L1 detection (paraffin specimens less than 2 years old or fresh tumor tissue)
7. patients with oropharyngeal carcinoma provide a test status for P16, using the IHC method.
8. Organ function levels must meet the following requirements (14 days prior to the first dose of study drug):

   Bone marrow:absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets (PLT) ≥ 100×109/L, hemoglobin (HB) ≥ 9g/dL (not transfused or receiving component blood within 14 days prior to testing); Liver: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal value (in case of liver metastases, AST and ALT ≤ 5 times the upper limit of normal value are allowed); serum creatinine ≤ 1.5 times the upper limit of normal value and endogenous creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula) Gault formula); International normalized ratio (INR), activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal (only for patients not receiving anticoagulation; patients receiving anticoagulation should keep anticoagulants within the therapeutically required range); Thyroid stimulating hormone (TSH) ≤ 1 x ULN (if abnormal FT3 and FT4 levels should be examined at the same time; if FT3 and FT4 levels are normal, the patient can be enrolled) Urine protein ≤ 1+, if urine protein > 1+, 24-hour urine protein measurement should be collected, and its total amount should be ≤ 1 gram; Normal cardiac function, i.e. normal or abnormal ECG examination without clinical significance and cardiac ultrasound showing left ventricular ejection fraction (LVEF) >50%.
9. female subjects of reproductive potential must have a negative serum pregnancy test prior to the first dose of the trial drug; 10. male or female subjects of reproductive potential must be using a highly effective method of contraception (e.g., oral contraceptive pills, intrauterine device, abstinence from sexual intercourse, or barrier method of contraception in combination with spermicide) throughout the trial and continue to use contraception for 90 days after the end of treatment.

11. Subjects voluntarily enrolled in the study, signed an informed consent form, were compliant and cooperative with follow-up.

Exclusion Criteria:

1. with distant metastatic lesions or localized lesions not indicated for surgery (patients with stage IVb or IVc)
2. have progressed within 6 months after systemic therapy directed at locally advanced squamous head and neck cancer.
3. a prior history of primary nasopharyngeal cancer tumor.
4. patients who have participated or are participating in a clinical trial of another drug/therapy within 4 weeks prior to the first dose of the study drug.
5. underwent/received major surgery or have not recovered from the side effects of such surgery, live vaccination, immunotherapy within 4 weeks prior to the first dosing of the study drug, and radiation therapy within 2 weeks.
6. receiving any other concurrent antitumor therapy.
7. the patient has any active autoimmune disease or a history of autoimmune disease (e.g., the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism; vitiligo that does not require systemic therapy may be included; asthma that has completely resolved in childhood and does not require any intervention in adulthood may be included; patients requiring bronchial (asthma that requires medical intervention with bronchodilators cannot be included).
8. patients who are on immunosuppressive, or systemic hormone therapy for immunosuppressive purposes (doses >10 mg/day of prednisone or other equipotent hormones) and continue to use them within 2 weeks prior to enrollment
9. a history of other malignancies within the past 5 years, with the exception of cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early stage prostate cancer and carcinoma in situ of the cervix
10. patients who have received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc., within 1 week prior to the first dose of the study drug
11. prior treatment with PD-1/PD-L1/PD-L2/CTLA-4 antibodies or activating or inhibitory agents targeting T-cell receptors (e.g., OX40, CD137)
12. prior drug treatment with cetuximab.
13. positive test results for HIV antibodies or syphilis spirochete antibodies
14. Patients with active hepatitis B or C:

    If HBsAg or HBcAb is positive, add HBV DNA test (the result is higher than the upper limit of the normal range).

    If HCV antibody test result is positive, add HCV RNA test (the result is higher than the upper limit of the normal range).
15. known to be allergic to recombinant humanized PD-1 monoclonal antibody drug and its components;
16. known to be allergic to EGFR monoclonal antibody drugs and their components;
17. have active lung disease (interstitial pneumonia, pneumonia, obstructive lung disease, asthma) or a history of active tuberculosis
18. have any uncontrollable clinical problem, including but not limited to: Persistent or active (severe) infection; Poorly medically controlled hypertension (blood pressure greater than 150/90 mmHg persistently).

    Poorly controlled diabetes mellitus; Cardiac disease (Class III/IV congestive heart failure or heart block as defined by the New York Heart Association);
19. the following conditions within 6 months prior to the first dose: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass graft; cerebrovascular accident, transient ischemic attack, cerebral embolism
20. having undergone stem cell transplantation or organ transplantation
21. persons with a history of psychotropic substance abuse that they are unable to abstain from or a history of psychiatric disorders
22. other serious, acute or chronic medical conditions or abnormalities in laboratory tests that, in the judgment of the investigator, may increase the risk associated with participation in the study, or may interfere with the interpretation of study results
23. Patients who, in the judgment of the investigator, have poor compliance or have other conditions that make them unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
One-year events-free survival rate | 12 months
  One-year EFS was defined as the percentage of participants without recurrence or death due to any cause at 12 month.

SECONDARY OUTCOMES:
disease-free survival | 12months
  DFS was defined as the time from salvage surgery to the earlier of recurrence or death due to any cause
overall survival | 12 months
  OS was defined as the time from salvage surgery to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
objective response rate | 24 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
major pathologic response | 24 months
  percentage of participants in the analysis population who have a tumor-active cell residue ≤10% in the surgical pathology specimens.
Participants Experiencing an Adverse Event (AE) | 12 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for treatment arm
Quality of life#EORTC QLQ-C30 scale# | 12 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, M.D., Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No